CLINICAL TRIAL: NCT03216629
Title: Sorry Not Sorry: Apologizing and Its Effect on Discomfort During Dressing Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Peng You, MD, London Health Sciences Centre
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 109333
Record Dates: First submitted 2017-07-11; First posted 2017-07-13 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Bandages; Pain; Empathy
Keywords: Pain; Empathy; Dressing change
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sorry (Experimental): A small strip of self-adhesive dressing (3cm by 4cm) will be applied to the back of the patients' participants' hand and side of neck. After one minute of acclimatization, the dressing will be removed by the examiner. During the removal, the examiner will say sorry repeatedly. Following the dressing removal, participant will rate their pain with a 10 point visual analog scale.
  Interventions: Behavioral: Saying "sorry"
- Not Sorry (No Intervention): A small strip of self-adhesive dressing (3cm by 4cm) will be applied to the back of the patients' participants' hand and side of neck. After one minute of acclimatization, the dressing will be removed by the examiner. During the removal, the examiner will remain silent. Following the dressing removal, participant will rate their pain with a 10 point visual analog scale.

INTERVENTIONS:
Behavioral: Saying "sorry" — The objective of this study is to investigate how empathy expressed in form of saying "sorry" affect the perception of pain during dressing change?
  Arms: Sorry

SUMMARY:
Use of dressing is common place following surgery, allowing for wounds to be covered and protected. Dressing material with adhesive contact layers or adhesive tape is integral to sealing off the wound. Mechanical stripping of stratum corneum during dressing removal causes pain and discomfort. During dressing removal, practitioners may at times apologize as a function of empathy. Previous study investigated speed of dressing removal and its effect on discomfort during dressing change. In this study, the investigators aim to investigate how empathy expressed in form of saying "sorry" affect the perception of pain during dressing change?

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers, age >18.

Exclusion Criteria:

* individuals with sensitivity to tape or dressing, anxiety disorders, or pain syndromes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Pain | Immediate
  Based on self reported 10 point visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Danielle MacNeil, MD, Principal Investigator — London Health Science Centre
Locations (1):
- London Health Science Centre - Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No